CLINICAL TRIAL: NCT03312816
Title: The Effect of Oxidized Plant Sterol Intake on Serum Concentrations of Plant Sterol Oxidation Products (POP)
Brief Title: Effect of Oxidized Plant Sterols on Serum Concentrations of Plant Sterol Oxidation Products (POP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FDS-SCC-2838
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 0 mg/d added POP
  Interventions: Other: cookies enriched with POP
- low dosage (Active Comparator): low added POP
  Interventions: Other: cookies enriched with POP
- Medium dose (Active Comparator): medium added POP
  Interventions: Other: cookies enriched with POP
- Hige dose (Active Comparator): high added POP
  Interventions: Other: cookies enriched with POP

INTERVENTIONS:
Other: cookies enriched with POP — Cookies

SUMMARY:
The study is a randomised, double-blind, placebocontrolled, parallel dose-response study with four study arms. Sixty subjects will be randomly allocated to consume study products containing varying amounts of plant sterol (PS) oxidation products (POP) or placebo for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women as judged by study physician.
* BMI > 18 and < 35 kg/m2.
* Total cholesterol levels at screening ≥5.0 and ≤8.0 mmol/L
* Blood pressure, heart rate, haematological and clinical chemical parameters within the normal reference range as judged by the study physician.

Exclusion Criteria:

* Recently (<6 months) diagnosed with cardiovascular event(s) (stroke, TIA (Transient ischemic attack), angina, myocardial infarction, heart failure), revascularization or systemic inflammatory conditions.
* Use of plant-sterol/stanol-enriched foods or supplements in the three months prior to the screening and/or during the study.
* Use of over-the-counter and prescribed medication which may interfere with study measurements (i.e. statins, ezetimibe, fibrates, diabetic drugs, angiotensin receptor blockers (ARB) and ACE (Angiotensin-converting enzyme) inhibitors)), to be judged by the principal investigator.
* Use of oral antibiotics (with the exception of topical antibiotics) in 40 days or less prior to Day -2.
* Pregnant or lactating women.
* Reported alcohol consumption > 14 units/week (female) or > 21 units/week (male).
* Reported intense sporting activities > 10 hours/week.
* Reported weight loss or gain of 3 kg or more during a period of 6 months prior to screening.
* Currently on a medically- or self-prescribed diet, or slimming diet, or the intention to use any kind of diet during the study.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months prior to screening and/or during the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
POP (plant sterol oxidation products) value | 0 to 42 days
  To estimate the change from baseline in serum POP concentration after intake of various POP doses.

SECONDARY OUTCOMES:
COP (cholesterol oxidation products) value | 0 to 42 days
  To estimate the change from baseline in serum COP concentrations after intake of various POP doses.
Ratio of serum POP concentration | 0 to 42 days
  To estimate the ratio of serum POP concentrations vs. COP concentrations after intake of various POP doses.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keicher, Dr, Principal Investigator — Charité Research Organisation GmbH
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany